CLINICAL TRIAL: NCT01764633
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study Assessing the Impact of Additional LDL-Cholesterol Reduction on Major Cardiovascular Events When Evolocumab (AMG 145) is Used in Combination With Statin Therapy In Patients With Clinically Evident Cardiovascular Disease
Brief Title: Further Cardiovascular Outcomes Research With PCSK9 Inhibition in Subjects With Elevated Risk
Acronym: FOURIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110118; 2014/01/004324 (Registry Identifier: Clinical Trials Registry- India (CTRI)); 2012-001398-97 (EudraCT Number)
Record Dates: First submitted 2013-01-08; First posted 2013-01-09 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Dyslipidemia
Keywords: High cholesterol; Treatment for high cholesterol; Lowering cholesterol; Lowering high cholesterol; Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections either once every 2 weeks (Q2W) or once a month (QM) according to their own preference.
  Interventions: Drug: Placebo
- Evolocumab (Experimental): Participants received evolocumab 140 mg Q2W or 420 mg QM subcutaneous injections according to their own preference.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered subcutaneously using a spring-based prefilled 1.0 mL autoinjector/pen.
  Other Names: AMG 145; Repatha
  Arms: Evolocumab
Drug: Placebo — Administered subcutaneously using a spring-based prefilled 1.0 mL autoinjector/pen.
  Arms: Placebo

SUMMARY:
The primary objective was to evaluate the effect of treatment with evolocumab, compared with placebo, on the risk for cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization, whichever occurs first, in patients with clinically evident cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 40 to ≤ 85 years of age
* History of clinically evident cardiovascular disease at high risk for a recurrent event
* Fasting low-density lipoprotein cholesterol (LDL-C) ≥ 70 mg/dL (≥ 1.8 mmol/L) ) or non-high-density lipoprotein cholesterol (non-HDL-C) ≥ 100 mg/dL (> 2.6 mmol/L)
* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L)

Exclusion Criteria:

* New York Heart Association (NYHA) class III or IV, or last known left ventricular ejection fraction < 30%
* Uncontrolled hypertension
* Uncontrolled or recurrent ventricular tachycardia
* Untreated hyperthyroidism or hypothyroidism
* Homozygous familial hypercholesterolemia
* LDL or plasma apheresis

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27564 (Actual)
Dates: Start 2013-02-08 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (978):
- United States (278):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Alhambra, California
  - Research Site, Banning, California
  - Research Site, Beverly Hills, California
  - Research Site, Encino, California
  - Research Site, Escondido, California
  - Research Site, Glendale, California
  - Research Site, Harbor City, California
  - Research Site, Huntington Beach, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Oceanside, California
  - Research Site, Oxnard, California
  - Research Site, Palm Springs, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Pedro, California
  - Research Site, Santa Ana, California
  - Research Site, Tarzana, California
  - Research Site, Thousand Oaks, California
  - Research Site, Torrance, California
  - Research Site, Valley Village, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Greeley, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Longmont, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Seaford, Delaware
  - Research Site, Wilmington, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlantis, Florida
  - Research Site, Aventura, Florida
  - Research Site, Bay Pines, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Fleming Island, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Largo, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Sanford, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Wellington, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, East Point, Georgia
  - Research Site, Eatonton, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Suwanee, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Nampa, Idaho
  - Research Site, Addison, Illinois
  - Research Site, Belleville, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, Jerseyville, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Des Moines, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Waterloo, Iowa
  - Research Site, Hutchinson, Kansas
  - Research Site, Kansas City, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Hammond, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Natchitoches, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Biddeford, Maine
  - Research Site, Portland, Maine
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Charlotte Hall, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Hollywood, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Ayer, Massachusetts
  - Research Site, Billerica, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Hyannis, Massachusetts
  - Research Site, Newton, Massachusetts
  - Research Site, Quincy, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Watertown, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Dearborn, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Grandville, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Novi, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Olive Branch, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Great Falls, Montana
  - Research Site, Kalispell, Montana
  - Research Site, Missoula, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Elizabeth, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Westwood, New Jersey
  - Research Site, Albany, New York
  - Research Site, Buffalo, New York
  - Research Site, Cortlandt Manor, New York
  - Research Site, Kingston, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Stony Brook, New York
  - Research Site, Syracuse, New York
  - Research Site, Troy, New York
  - Research Site, West Seneca, New York
  - Research Site, Williamsville, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Calabash, North Carolina
  - Research Site, Cary, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Grand Forks, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Elyria, Ohio
  - Research Site, Garfield Heights, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Westlake, Ohio
  - Research Site, Willoughby, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Pryor, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Altoona, Pennsylvania
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Chambersburg, Pennsylvania
  - Research Site, Feasterville, Pennsylvania
  - Research Site, Indiana, Pennsylvania
  - Research Site, Jersey Shore, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Cranston, Rhode Island
  - Research Site, Cumberland, Rhode Island
  - Research Site, Johnston, Rhode Island
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Fountain Inn, South Carolina
  - Research Site, Moncks Corner, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, North Myrtle Beach, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Germantown, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Grapevine, Texas
  - Research Site, Houston, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Longview, Texas
  - Research Site, Odessa, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Tomball, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Layton, Utah
  - Research Site, Murray, Utah
  - Research Site, West Jordan, Utah
  - Research Site, White River Junction, Vermont
  - Research Site, Burke, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Hopewell, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Federal Way, Washington
  - Research Site, Seattle, Washington
  - Research Site, Selah, Washington
  - Research Site, Green Bay, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Marshfield, Wisconsin
- Argentina (11):
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, La Plata, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Salta
- Australia (20):
  - Research Site, Woden, Australian Capital Territory
  - Research Site, Camperdown, New South Wales
  - Research Site, Concord, New South Wales
  - Research Site, Kogarah, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, Woolloongabba, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research Site, Herston, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Ashford, South Australia
  - Research Site, Fullarton, South Australia
  - Research Site, Woodville South, South Australia
  - Research Site, Hobart, Tasmania
  - Research Site, Box Hill, Victoria
  - Research Site, Epping, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Nedlands, Western Australia
- Austria (6):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (13):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Blankenberge
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Gozée
  - Research Site, Ieper
  - Research Site, La Louvière
  - Research Site, Liège
  - Research Site, Lodelinsart
  - Research Site, Natoye
  - Research Site, Turnhout
- Brazil (15):
  - Research Site, Fortaleza, Ceará
  - Research Site, Vitória, Espírito Santo
  - Research Site, Brasília, Federal District
  - Research Site, Goiânia, Goiás
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Campina Grande do Sul, Paraná
  - Research Site, Curitiba, Paraná
  - Research Site, Canoas, Rio Grande do Sul
  - Research Site, Passo Fundo, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Campinas, São Paulo
  - Research Site, São José do Rio Preto, São Paulo
  - Research Site, São Paulo, São Paulo
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (7):
  - Research Site, Haskovo
  - Research Site, Kazanlak
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (34):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Strathroy, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Granby, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Lachine, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Westmout, Quebec
  - Research Site, Regina, Saskatchewan
- Chile (3):
  - Research Site, Temuco, Cautín
  - Research Site, Osorno
  - Research Site, Santiago
- China (29):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Harbin, Heilongjiang
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changde, Hunan
  - Research Site, Changsha, Hunan
  - Research Site, Xiangtan, Hunan
  - Research Site, Zhuzhou, Hunan
  - Research Site, Baotou, Inner Mongolia
  - Research Site, Hohhot, Inner Mongolia
  - Research Site, Suzhou, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Xuzhou, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Siping, Jilin
  - Research Site, Dalian, Liaoning
  - Research Site, Shenyang, Liaoning
  - Research Site, Yinchuan, Ningxia
  - Research Site, Qingdao, Shandong
  - Research Site, Taiyuan, Shanxi
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Ürümqi, Xinjiang
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Linhai, Zhejiang
  - Research Site, Ningbo, Zhejiang
  - Research Site, Wenzhou, Zhejiang
  - Research Site, Beijing
  - Research Site, Tianjin
- Colombia (8):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Manizales, Caldas Department
  - Research Site, Bogota, Cundinamarca
  - Research Site, Cartagena, Departamento de Bolívar
  - Research Site, Armenia, Quindío Department
  - Research Site, Floridablanca, Santander Department
  - Research Site, Cali, Valle del Cauca Department
- Czechia (41):
  - Research Site, Benátky nad Jizerou
  - Research Site, Benešov
  - Research Site, Beroun
  - Research Site, Bílovec
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, České Budějovice
  - Research Site, Český Krumlov
  - Research Site, Havlíčkův Brod
  - Research Site, Hodonín
  - Research Site, Hradec Králové
  - Research Site, Hranice
  - Research Site, Jihlava
  - Research Site, Kladno
  - Research Site, Klatovy IV
  - Research Site, Kutná Hora
  - Research Site, Liberec
  - Research Site, Litoměřice
  - Research Site, Litomyšl
  - Research Site, Milevsko
  - Research Site, Mladá Boleslav
  - Research Site, Mohelnice
  - Research Site, Moravské Budějovice
  - Research Site, Nymburk
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Ostrava-Poruba
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Polička
  - Research Site, Prachatice
  - Research Site, Prague
  - Research Site, Praha 5 - Smichov
  - Research Site, Pribram VIII
  - Research Site, Přerov
  - Research Site, Svitavy
  - Research Site, Teplice
  - Research Site, Uherské Hradiště
  - Research Site, Zábřeh nad Odrou
  - Research Site, Znojmo
- Denmark (14):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Ballerup Municipality
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Glostrup Municipality
  - Research Site, Hvidovre
  - Research Site, København S
  - Research Site, Køge
  - Research Site, Odense
  - Research Site, Roskilde
  - Research Site, Svendborg
  - Research Site, Vejle
  - Research Site, Viborg
- Estonia (3):
  - Research Site, Harjumaa
  - Research Site, Paide
  - Research Site, Tallinn
- Finland (8):
  - Research Site, Hämeenlinna
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Kokkola
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Tampere
  - Research Site, Turku
- France (28):
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Chambray-lès-Tours
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Le Coudray
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Metz
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vesoul
- Germany (28):
  - Research Site, Bad Krozingen
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Demmin
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Frankfurt am Main
  - Research Site, Giessen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Ingelheim
  - Research Site, Kassel
  - Research Site, Lahr
  - Research Site, Leipzig
  - Research Site, Limburg
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Stuttgart
  - Research Site, Ulm
  - Research Site, Witten
  - Research Site, Wuppertal
- Greece (10):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Chalcis
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Nikaia, Piraeus
  - Research Site, Piraeus
  - Research Site, Rhodes
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (18):
  - Research Site, Balatonfüred
  - Research Site, Berettyóújfalu
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Gyöngyös
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Komárom
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg
- Iceland (2):
  - Research Site, Kopavogur
  - Research Site, Reykjavik
- India (12):
  - Research Site, Vijayawada, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Gurgaon, Haryana
  - Research Site, Belagavi, Karnataka
  - Research Site, Mysore, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Kolkata, West Bengal
- Ireland (3):
  - Research Site, Ballinasloe
  - Research Site, Dublin
  - Research Site, Galway
- Israel (10):
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Herzliya-on-sea
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Netanya
  - Research Site, Rehovot
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (18):
  - Research Site, Ascoli Piceno
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Chieti
  - Research Site, Colleferro RM
  - Research Site, Cortona AR
  - Research Site, Florence
  - Research Site, L’Aquila
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Sanremo (IM)
  - Research Site, Siena
- Japan (55):
  - Research Site, Ichinomiya-shi, Aichi-ken
  - Research Site, Kasugai-shi, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Toyohashi, Aichi-ken
  - Research Site, Chiba, Chiba
  - Research Site, Matsudo-shi, Chiba
  - Research Site, Niihama-shi, Ehime
  - Research Site, Saijo-shi, Ehime
  - Research Site, Chikushi-gun, Fukuoka
  - Research Site, Chikushino-shi, Fukuoka
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Itoshima-shi, Fukuoka
  - Research Site, Koga-shi, Fukuoka
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Okawa-shi, Fukuoka
  - Research Site, Koriyama-shi, Fukushima
  - Research Site, Kure-shi, Hiroshima
  - Research Site, Otake-shi, Hiroshima
  - Research Site, Asahikawa-shi, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Himeji-shi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Toride-shi, Ibaraki
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Sanuki-shi, Kagawa-ken
  - Research Site, Fujisawa-shi, Kanagawa
  - Research Site, Odawara-shi, Kanagawa
  - Research Site, Sagamihara-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Higashisonogi-gun, Nagasaki
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Omura-shi, Nagasaki
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Okayama, Okayama-ken
  - Research Site, Okinawa-shi, Okinawa
  - Research Site, Shimajiri-gun, Okinawa
  - Research Site, Urasoe-shi, Okinawa
  - Research Site, Osaka, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Kawaguchi-shi, Saitama
  - Research Site, Kusatsu-shi, Shiga
  - Research Site, Hamada-shi, Shimane
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Komatsushima-shi, Tokushima
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Musashimurayama-shi, Tokyo
  - Research Site, Tachikawa-shi, Tokyo
  - Research Site, Chuo-shi, Yamanashi
- Latvia (5):
  - Research Site, Daugavpils
  - Research Site, Kuldīga
  - Research Site, Liepāja
  - Research Site, Ogre
  - Research Site, Riga
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Vilnius
- Malaysia (7):
  - Research Site, Johor Bahru, Johor
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Taiping, Perak
  - Research Site, Kota Kinabalu, Sabah
  - Research Site, George Town
  - Research Site, Kuala Lumpur
  - Research Site, Malacca
- Mexico (12):
  - Research Site, Torreón, Coahuila
  - Research Site, León, Guanajuato
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, Querétaro City, Querétaro
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Culiacán, Sinaloa
  - Research Site, Tampico, Tamaulipas
  - Research Site, Xalapa, Veracruz
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
- Netherlands (29):
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Amstelveen
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Beverwijk
  - Research Site, Den Helder
  - Research Site, Deventer
  - Research Site, Doetinchem
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Goes
  - Research Site, Gorinchem
  - Research Site, Gouda
  - Research Site, Harderwijk
  - Research Site, Helmond
  - Research Site, Hoogeveen
  - Research Site, Hoorn
  - Research Site, Leiden
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Purmerend
  - Research Site, Rotterdam
  - Research Site, Sneek
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Uden
  - Research Site, Veldhoven
  - Research Site, Venlo
- New Zealand (3):
  - Research Site, Christchurch
  - Research Site, Papatoetoe, Auckland
  - Research Site, Tauranga
- Norway (9):
  - Research Site, Ålesund
  - Research Site, Bekkestua
  - Research Site, Bodø
  - Research Site, Hamar
  - Research Site, Lierskogen
  - Research Site, Oslo
  - Research Site, Skedsmokorset
  - Research Site, Skien
  - Research Site, Stavanger
- Philippines (9):
  - Research Site, Davao City, Davao Region
  - Research Site, Angeles
  - Research Site, Baguio City
  - Research Site, Dasmariñas Cavite
  - Research Site, Iloilo City
  - Research Site, Makati City
  - Research Site, Manila
  - Research Site, Marikiina
  - Research Site, Quezon City
- Poland (29):
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Giżycko
  - Research Site, Jelenia Góra
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Nowa Sól
  - Research Site, Nysa
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Pszczyna
  - Research Site, Puławy
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Skierniewice
  - Research Site, Starogard Gdański
  - Research Site, Staszów
  - Research Site, Świdnik
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Zamość
- Portugal (8):
  - Research Site, Almada
  - Research Site, Amadora
  - Research Site, Carnaxide
  - Research Site, Coimbra
  - Research Site, Covilha
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Setúbal
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Timișoara
- Russia (15):
  - Research Site, Barnaul
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kemerovo
  - Research Site, Kirov
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Pushkin
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tomsk
  - Research Site, Tyumen
  - Research Site, Yekaterinburg
- Research Site, Singapore, Singapore
- Slovakia (18):
  - Research Site, Bardejov
  - Research Site, Bánovce nad Bebravou
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Dolný Kubín
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Martin
  - Research Site, Moldava nad Bodvou
  - Research Site, Nitra
  - Research Site, Nové Zámky
  - Research Site, Prešov
  - Research Site, Rimavská Sobota
  - Research Site, Rožňava
  - Research Site, Snina
  - Research Site, Svidník
  - Research Site, Trenčín
  - Research Site, Trnava
- South Africa (21):
  - Research Site, Port Elizabeth, Eastern Cape
  - Research Site, Bloemfontein, Free State
  - Research Site, Alberton, Gauteng
  - Research Site, Boksburg, Gauteng
  - Research Site, Centurion, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Midrand, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Pretoria West, Gauteng
  - Research Site, Soweto, Gauteng
  - Research Site, Sunninghill, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, eManzimtoti, KwaZulu-Natal
  - Research Site, Tongaat, KwaZulu-Natal
  - Research Site, Kuils River, Western Cape
  - Research Site, Paarl, Western Cape
  - Research Site, Parow, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Worcester, Western Cape
  - Research Site, Cape Town
  - Research Site, Kempton Park
- South Korea (7):
  - Research Site, Busan, Seo-gu
  - Research Site, Daejeon
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Gwangju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (11):
  - Research Site, Almería, Andalusia
  - Research Site, Córdoba, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, Galdakao, Basque Country
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Vigo, Galicia
  - Research Site, El Palmar, Murcia
  - Research Site, Sant Joan d'Alacant, Valencia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Sweden (15):
  - Research Site, Bollnäs
  - Research Site, Eksjö
  - Research Site, Eskilstuna
  - Research Site, Falun
  - Research Site, Helsingborg
  - Research Site, Jönköping
  - Research Site, Linköping
  - Research Site, Luleå
  - Research Site, Lund
  - Research Site, Örebro
  - Research Site, Östersund
  - Research Site, Stockholm
  - Research Site, Uddevalla
  - Research Site, Umeå
  - Research Site, Västerås
- Switzerland (9):
  - Research Site, Baden
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Lugano
  - Research Site, Sion
  - Research Site, Winterthur
  - Research Site, Zurich
- Taiwan (7):
  - Research Site, New Taipei City, Taipei
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Turkey (Türkiye) (7):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Konya
  - Research Site, Sivas
- Ukraine (9):
  - Research Site, Cherkasy
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Luhansk
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zaporizhzhya
- United Kingdom (62):
  - Research Site, Aberdeen
  - Research Site, Addlestone
  - Research Site, Arnsley
  - Research Site, Basildon
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Bournemouth
  - Research Site, Bury St Edmunds
  - Research Site, Canterbury
  - Research Site, Cardiff
  - Research Site, Chesterfield
  - Research Site, Chippenham
  - Research Site, Chorley
  - Research Site, Colchester
  - Research Site, Cottingham
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Haxey, Doncaster
  - Research Site, Hayle
  - Research Site, Hexham
  - Research Site, Hitchin
  - Research Site, Inverness
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Luton
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral
  - Research Site, Middlesbrough
  - Research Site, Newport
  - Research Site, Northampton
  - Research Site, Nottingham
  - Research Site, Nuneaton
  - Research Site, Penzance
  - Research Site, Plymouth
  - Research Site, Portsmouth
  - Research Site, Reading
  - Research Site, Rotherham
  - Research Site, Royal Leamington Spa
  - Research Site, Rugby
  - Research Site, Saint Leonards-on-Sea
  - Research Site, Sandbach
  - Research Site, Sheffield
  - Research Site, St Austell
  - Research Site, Stevenage
  - Research Site, Stoke-on-Trent
  - Research Site, Swansea
  - Research Site, Telford
  - Research Site, Torquay
  - Research Site, Welwyn Garden City
  - Research Site, West Bromwich
  - Research Site, Whitby
  - Research Site, Wiltshire
  - Research Site, Wolverhampton
  - Research Site, Worcester
  - Research Site, Wrexham
  - Research Site, York

REFERENCES:
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Fonarow GC, Keech AC, Pedersen TR, Giugliano RP, Sever PS, Lindgren P, van Hout B, Villa G, Qian Y, Somaratne R, Sabatine MS. Cost-effectiveness of Evolocumab Therapy for Reducing Cardiovascular Events in Patients With Atherosclerotic Cardiovascular Disease. JAMA Cardiol. 2017 Oct 1;2(10):1069-1078. doi: 10.1001/jamacardio.2017.2762. PMID 28832867
- [Background] Fonarow GC, van Hout B, Villa G, Arellano J, Lindgren P. Updated Cost-effectiveness Analysis of Evolocumab in Patients With Very High-risk Atherosclerotic Cardiovascular Disease. JAMA Cardiol. 2019 Jul 1;4(7):691-695. doi: 10.1001/jamacardio.2019.1647. PMID 31166576
- [Background] Schludi B, Giugliano RP, Sabatine MS, Raal FJ, Teramoto T, Koren MJ, Stein EA, Wang H, Monsalvo ML. Time-averaged low-density lipoprotein cholesterol lowering with evolocumab: Pooled analysis of phase 2 trials. J Clin Lipidol. 2022 Jul-Aug;16(4):538-543. doi: 10.1016/j.jacl.2022.05.069. Epub 2022 Jun 6. PMID 35760720
- [Background] Berg DD, Moura FA, Bellavia A, Scirica BM, Wiviott SD, Bhatt DL, Raz I, Bohula EA, Giugliano RP, Park JG, Feinberg MW, Braunwald E, Morrow DA, Sabatine MS. Assessment of Atherothrombotic Risk in Patients With Type 2 Diabetes Mellitus. J Am Coll Cardiol. 2023 Jun 27;81(25):2391-2402. doi: 10.1016/j.jacc.2023.04.031. PMID 37344040
- [Background] Clinical Benefit of Evolocumab Treatment Among Patients With Atherosclerotic Cardiovascular Disease: Exploration Based on the Chinese Subgroup of FOURIER Study, ZHANG Lihua1 , LI Weimin2 , YAO Zhuhua3 , CHEN Jiyan4 , DONG Jun5 , LI Jing1 (Chinese Circulation Journal, 2023, 38: 704.)
- [Derived] Monguillon V, Kelly PJ, O'Donoghue ML, Park JG, Bohula EA, Saver JL, Atar D, Keech AC, Sever PS, Wang H, Paiva da Silva Lima G, Sabatine MS, Giugliano RP. Efficacy and Safety of Very Low Achieved LDL Cholesterol in Patients With Previous Ischemic Stroke. Circulation. 2026 Jan 13;153(2):86-93. doi: 10.1161/CIRCULATIONAHA.125.077549. Epub 2025 Nov 3. PMID 41178569
- [Derived] Zimerman A, Kunzler ALF, Weber BN, Ran X, Murphy SA, Wang H, Honarpour N, Keech AC, Sever PS, Sabatine MS, Giugliano RP. Intensive Lowering of LDL Cholesterol Levels With Evolocumab in Autoimmune or Inflammatory Diseases: An Analysis of the FOURIER Trial. Circulation. 2025 May 20;151(20):1467-1476. doi: 10.1161/CIRCULATIONAHA.124.072756. Epub 2025 Apr 21. PMID 40255182
- [Derived] Gaba P, O'Donoghue ML, Park JG, Wiviott SD, Atar D, Kuder JF, Im K, Murphy SA, De Ferrari GM, Gaciong ZA, Toth K, Gouni-Berthold I, Lopez-Miranda J, Schiele F, Mach F, Flores-Arredondo JH, Lopez JAG, Elliott-Davey M, Wang B, Monsalvo ML, Abbasi S, Giugliano RP, Sabatine MS. Association Between Achieved Low-Density Lipoprotein Cholesterol Levels and Long-Term Cardiovascular and Safety Outcomes: An Analysis of FOURIER-OLE. Circulation. 2023 Apr 18;147(16):1192-1203. doi: 10.1161/CIRCULATIONAHA.122.063399. Epub 2023 Feb 13. PMID 36779348
- [Derived] Erviti J, Wright J, Bassett K, Ben-Eltriki M, Jauca C, Saiz LC, Leache L, Gutierrez-Valencia M, Perry TL. Restoring mortality data in the FOURIER cardiovascular outcomes trial of evolocumab in patients with cardiovascular disease: a reanalysis based on regulatory data. BMJ Open. 2022 Dec 30;12(12):e060172. doi: 10.1136/bmjopen-2021-060172. PMID 36585131
- [Derived] Fagundes A Jr, Morrow DA, Oyama K, Furtado RHM, Zelniker TA, Tang M, Kuder JF, Murphy SA, Hamer A, Keech AC, Sever P, Giugliano RP, Sabatine MS, Bergmark BA. Biomarker Prediction of Complex Coronary Revascularization Procedures in the FOURIER Trial. J Am Coll Cardiol. 2022 Aug 30;80(9):887-897. doi: 10.1016/j.jacc.2022.05.051. PMID 36007987
- [Derived] Furtado RHM, Fagundes AA Jr, Oyama K, Zelniker TA, Tang M, Kuder JF, Murphy SA, Hamer A, Wang H, Keech AC, Giugliano RP, Sabatine MS, Bergmark BA. Effect of Evolocumab in Patients With Prior Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2022 Mar;15(3):e011382. doi: 10.1161/CIRCINTERVENTIONS.121.011382. Epub 2022 Feb 25. PMID 35209731
- [Derived] Oyama K, Giugliano RP, Tang M, Bonaca MP, Saver JL, Murphy SA, Ruzza A, Keech AC, Sever PS, Sabatine MS, Bergmark BA. Effect of evolocumab on acute arterial events across all vascular territories : results from the FOURIER trial. Eur Heart J. 2021 Dec 14;42(47):4821-4829. doi: 10.1093/eurheartj/ehab604. PMID 34537830
- [Derived] Keech AC, Oyama K, Sever PS, Tang M, Murphy SA, Hirayama A, Lu C, Tay L, Deedwania PC, Siu CW, Lira Pineda A, Choi D, Charng MJ, Amerena J, Wan Ahmad WA, Chopra VK, Pedersen TR, Giugliano RP, Sabatine MS; FOURIER Study Group. Efficacy and Safety of Long-Term Evolocumab Use Among Asian Subjects - A Subgroup Analysis of the Further Cardiovascular Outcomes Research With PCSK9 Inhibition in Subjects With Elevated Risk (FOURIER) Trial. Circ J. 2021 Oct 25;85(11):2063-2070. doi: 10.1253/circj.CJ-20-1051. Epub 2021 May 15. PMID 33980763
- [Derived] Oyama K, Furtado RHM, Fagundes A Jr, Zelniker TA, Tang M, Kuder J, Murphy SA, Hamer A, Wang H, Keech AC, Giugliano RP, Sabatine MS, Bergmark BA. Effect of Evolocumab on Complex Coronary Disease Requiring Revascularization. J Am Coll Cardiol. 2021 Jan 26;77(3):259-267. doi: 10.1016/j.jacc.2020.11.011. Epub 2020 Nov 13. PMID 33197560
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Deedwania P, Murphy SA, Scheen A, Badariene J, Pineda AL, Honarpour N, Keech AC, Sever PS, Pedersen TR, Sabatine MS, Giugliano RP. Efficacy and Safety of PCSK9 Inhibition With Evolocumab in Reducing Cardiovascular Events in Patients With Metabolic Syndrome Receiving Statin Therapy: Secondary Analysis From the FOURIER Randomized Clinical Trial. JAMA Cardiol. 2021 Feb 1;6(2):139-147. doi: 10.1001/jamacardio.2020.3151. PMID 32785614
- [Derived] Gencer B, Mach F, Murphy SA, De Ferrari GM, Huber K, Lewis BS, Ferreira J, Kurtz CE, Wang H, Honarpour N, Keech AC, Sever PS, Pedersen TR, Sabatine MS, Giugliano RP. Efficacy of Evolocumab on Cardiovascular Outcomes in Patients With Recent Myocardial Infarction: A Prespecified Secondary Analysis From the FOURIER Trial. JAMA Cardiol. 2020 Aug 1;5(8):952-957. doi: 10.1001/jamacardio.2020.0882. PMID 32432684
- [Derived] Bergmark BA, O'Donoghue ML, Murphy SA, Kuder JF, Ezhov MV, Ceska R, Gouni-Berthold I, Jensen HK, Tokgozoglu SL, Mach F, Huber K, Gaciong Z, Lewis BS, Schiele F, Jukema JW, Pedersen TR, Giugliano RP, Sabatine MS. An Exploratory Analysis of Proprotein Convertase Subtilisin/Kexin Type 9 Inhibition and Aortic Stenosis in the FOURIER Trial. JAMA Cardiol. 2020 Jun 1;5(6):709-713. doi: 10.1001/jamacardio.2020.0728. PMID 32347887
- [Derived] Wiviott SD, Giugliano RP, Morrow DA, De Ferrari GM, Lewis BS, Huber K, Kuder JF, Murphy SA, Forni DM, Kurtz CE, Honarpour N, Keech AC, Sever PS, Pedersen TR, Sabatine MS. Effect of Evolocumab on Type and Size of Subsequent Myocardial Infarction: A Prespecified Analysis of the FOURIER Randomized Clinical Trial. JAMA Cardiol. 2020 Jul 1;5(7):787-793. doi: 10.1001/jamacardio.2020.0764. PMID 32347885
- [Derived] Giugliano RP, Pedersen TR, Saver JL, Sever PS, Keech AC, Bohula EA, Murphy SA, Wasserman SM, Honarpour N, Wang H, Lira Pineda A, Sabatine MS; FOURIER Investigators. Stroke Prevention With the PCSK9 (Proprotein Convertase Subtilisin-Kexin Type 9) Inhibitor Evolocumab Added to Statin in High-Risk Patients With Stable Atherosclerosis. Stroke. 2020 May;51(5):1546-1554. doi: 10.1161/STROKEAHA.119.027759. Epub 2020 Apr 21. PMID 32312223
- [Derived] Charytan DM, Sabatine MS, Pedersen TR, Im K, Park JG, Pineda AL, Wasserman SM, Deedwania P, Olsson AG, Sever PS, Keech AC, Giugliano RP; FOURIER Steering Committee and Investigators. Efficacy and Safety of Evolocumab in Chronic Kidney Disease in the FOURIER Trial. J Am Coll Cardiol. 2019 Jun 18;73(23):2961-2970. doi: 10.1016/j.jacc.2019.03.513. PMID 31196453
- [Derived] Murphy SA, Pedersen TR, Gaciong ZA, Ceska R, Ezhov MV, Connolly DL, Jukema JW, Toth K, Tikkanen MJ, Im K, Wiviott SD, Kurtz CE, Honarpour N, Giugliano RP, Keech AC, Sever PS, Sabatine MS. Effect of the PCSK9 Inhibitor Evolocumab on Total Cardiovascular Events in Patients With Cardiovascular Disease: A Prespecified Analysis From the FOURIER Trial. JAMA Cardiol. 2019 Jul 1;4(7):613-619. doi: 10.1001/jamacardio.2019.0886. PMID 31116355
- [Derived] O'Donoghue ML, Fazio S, Giugliano RP, Stroes ESG, Kanevsky E, Gouni-Berthold I, Im K, Lira Pineda A, Wasserman SM, Ceska R, Ezhov MV, Jukema JW, Jensen HK, Tokgozoglu SL, Mach F, Huber K, Sever PS, Keech AC, Pedersen TR, Sabatine MS. Lipoprotein(a), PCSK9 Inhibition, and Cardiovascular Risk. Circulation. 2019 Mar 19;139(12):1483-1492. doi: 10.1161/CIRCULATIONAHA.118.037184. PMID 30586750
- [Derived] Qamar A, Giugliano RP, Keech AC, Kuder JF, Murphy SA, Kurtz CE, Wasserman SM, Sever PS, Pedersen TR, Sabatine MS. Interindividual Variation in Low-Density Lipoprotein Cholesterol Level Reduction With Evolocumab: An Analysis of FOURIER Trial Data. JAMA Cardiol. 2019 Jan 1;4(1):59-63. doi: 10.1001/jamacardio.2018.4178. PMID 30540337
- [Derived] Martin SS, Giugliano RP, Murphy SA, Wasserman SM, Stein EA, Ceska R, Lopez-Miranda J, Georgiev B, Lorenzatti AJ, Tikkanen MJ, Sever PS, Keech AC, Pedersen TR, Sabatine MS. Comparison of Low-Density Lipoprotein Cholesterol Assessment by Martin/Hopkins Estimation, Friedewald Estimation, and Preparative Ultracentrifugation: Insights From the FOURIER Trial. JAMA Cardiol. 2018 Aug 1;3(8):749-753. doi: 10.1001/jamacardio.2018.1533. PMID 29898218
- [Derived] Sabatine MS, De Ferrari GM, Giugliano RP, Huber K, Lewis BS, Ferreira J, Kuder JF, Murphy SA, Wiviott SD, Kurtz CE, Honarpour N, Keech AC, Sever PS, Pedersen TR. Clinical Benefit of Evolocumab by Severity and Extent of Coronary Artery Disease: Analysis From FOURIER. Circulation. 2018 Aug 21;138(8):756-766. doi: 10.1161/CIRCULATIONAHA.118.034309. PMID 29626068
- [Derived] Bohula EA, Giugliano RP, Leiter LA, Verma S, Park JG, Sever PS, Lira Pineda A, Honarpour N, Wang H, Murphy SA, Keech A, Pedersen TR, Sabatine MS. Inflammatory and Cholesterol Risk in the FOURIER Trial. Circulation. 2018 Jul 10;138(2):131-140. doi: 10.1161/CIRCULATIONAHA.118.034032. Epub 2018 Mar 12. PMID 29530884
- [Derived] Bonaca MP, Nault P, Giugliano RP, Keech AC, Pineda AL, Kanevsky E, Kuder J, Murphy SA, Jukema JW, Lewis BS, Tokgozoglu L, Somaratne R, Sever PS, Pedersen TR, Sabatine MS. Low-Density Lipoprotein Cholesterol Lowering With Evolocumab and Outcomes in Patients With Peripheral Artery Disease: Insights From the FOURIER Trial (Further Cardiovascular Outcomes Research With PCSK9 Inhibition in Subjects With Elevated Risk). Circulation. 2018 Jan 23;137(4):338-350. doi: 10.1161/CIRCULATIONAHA.117.032235. Epub 2017 Nov 13. PMID 29133605
- [Derived] Sabatine MS, Leiter LA, Wiviott SD, Giugliano RP, Deedwania P, De Ferrari GM, Murphy SA, Kuder JF, Gouni-Berthold I, Lewis BS, Handelsman Y, Pineda AL, Honarpour N, Keech AC, Sever PS, Pedersen TR. Cardiovascular safety and efficacy of the PCSK9 inhibitor evolocumab in patients with and without diabetes and the effect of evolocumab on glycaemia and risk of new-onset diabetes: a prespecified analysis of the FOURIER randomised controlled trial. Lancet Diabetes Endocrinol. 2017 Dec;5(12):941-950. doi: 10.1016/S2213-8587(17)30313-3. Epub 2017 Sep 15. PMID 28927706
- [Derived] Giugliano RP, Pedersen TR, Park JG, De Ferrari GM, Gaciong ZA, Ceska R, Toth K, Gouni-Berthold I, Lopez-Miranda J, Schiele F, Mach F, Ott BR, Kanevsky E, Pineda AL, Somaratne R, Wasserman SM, Keech AC, Sever PS, Sabatine MS; FOURIER Investigators. Clinical efficacy and safety of achieving very low LDL-cholesterol concentrations with the PCSK9 inhibitor evolocumab: a prespecified secondary analysis of the FOURIER trial. Lancet. 2017 Oct 28;390(10106):1962-1971. doi: 10.1016/S0140-6736(17)32290-0. Epub 2017 Aug 28. PMID 28859947
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1242 clinical centers in 49 countries in the regions of Europe (62.9%), North America (16.6%), Asia Pacific (13.9%), and Latin America (6.6%) from 08 February 2013 to 05 June 2015.
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to receive either subcutaneous (SC) evolocumab or placebo. Randomization was stratified by the final screening low-density lipoprotein cholesterol (LDL-C) level (< 85 mg/dL vs ≥ 85 mg/dL) and by geographical region.
Groups:
- Evolocumab: Participants received evolocumab subcutaneous injections either 140 mg Q2W or 420 mg QM according to their own preference.
Period: Overall Study
Arm/Group | Placebo | Evolocumab
Started | 13780 | 13784
Received Treatment | 13756 | 13769
Completed | 13662 | 13691
Not Completed | 118 | 93
Not completed — Withdrawal by Subject | 105 | 88
Not completed — Lost to Follow-up | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab | Total
Number analyzed (Participants) | 13780 | 13784 | 27564
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (8.9) | 62.5 (9.1) | 62.5 (9.0)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 7687 | 7623 | 15310
  ≥ 65 years | 6093 | 6161 | 12254
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3382 | 3387 | 6769
  Male | 10398 | 10397 | 20795
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1084 | 1093 | 2177
  Not Hispanic or Latino | 12694 | 12688 | 25382
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 80 | 60 | 140
  Asian | 1349 | 1374 | 2723
  Black or African American | 352 | 317 | 669
  Native Hawaiian or Other Pacific Islander | 11 | 15 | 26
  White | 11710 | 11748 | 23458
  Multiple | 12 | 19 | 31
  Other | 266 | 251 | 517
Low-density Lipoprotein Cholesterol [Count of Participants; unit: Participants]
  < 85 mg/dL | 4803 | 4809 | 9612
  ≥ 85 mg/dL | 8977 | 8975 | 17952
Geographical Region [Count of Participants; unit: Participants]
  Europe | 8669 | 8667 | 17336
  North America | 2284 | 2286 | 4570
  Latin America | 910 | 913 | 1823
  Asia Pacific | 1917 | 1918 | 3835

OUTCOME MEASURES:

1. Primary Outcome: Time to Cardiovascular Death, Myocardial Infarction, Hospitalization for Unstable Angina, Stroke, or Coronary Revascularization
Description: All deaths and potential endpoint events were adjudicated by an independent external Clinical Events Committee (CEC) led by the Thrombolysis in Myocardial Infarction (TIMI) Study Group, using standardized definitions based on the "Standardized Definitions for Cardiovascular and Stroke End Point Events in Clinical Trials and the Third Universal Definition of Myocardial Infarction".
  Time to cardiovascular death, myocardial infarction, stroke, hospitalization for unstable angina, or coronary revascularization was defined as the time from randomization to the first occurrence of any component of the composite endpoint and was analyzed using Kaplan-Meier (KM) survival analysis. KM estimates of the percentage of participants with an event are reported. Participants with no event were censored based on last non-fatal potential endpoint collection date.
Time Frame: Events that occurred from randomization to the last confirmed survival status date; the median duration of follow-up was 26 months. KM estimates at 6, 12, 18, 24, 30 and 36 months are reported.
Population: All randomized participants; The number of participants entered at each time point represents the number of participants at risk.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13276 | 13349
  KM estimate at 6 months | 3.11 [2.82 to 3.40] | 2.74 [2.47 to 3.01]
  KM estimate at 12 months: number analyzed (Participants) | 12822 | 12937
  KM estimate at 12 months | 6.01 [5.61 to 6.41] | 5.31 [4.93 to 5.68]
  KM estimate at 18 months: number analyzed (Participants) | 11837 | 12034
  KM estimate at 18 months | 8.32 [7.86 to 8.78] | 7.25 [6.81 to 7.68]
  KM estimate at 24 months: number analyzed (Participants) | 7589 | 7743
  KM estimate at 24 months | 10.66 [10.12 to 11.19] | 9.13 [8.63 to 9.63]
  KM estimate at 30 months: number analyzed (Participants) | 3589 | 3652
  KM estimate at 30 months | 12.72 [12.08 to 13.35] | 10.91 [10.31 to 11.50]
  KM estimate at 36 months: number analyzed (Participants) | 672 | 681
  KM estimate at 36 months | 14.64 [13.76 to 15.50] | 12.57 [11.70 to 13.42]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; The primary endpoint was compared between treatment groups at a significance level of 0.05; Test type: Superiority; p < 0.0001, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.79 to 0.92] — Based on a Cox model stratified by the randomization stratification factors

2. Secondary Outcome: Time to Cardiovascular Death, Myocardial Infarction, or Stroke
Description: All deaths and potential endpoint events were adjudicated by an independent external CEC led by the TIMI Study Group, using standardized definitions based on the "Standardized Definitions for Cardiovascular and Stroke End Point Events in Clinical Trials and the Third Universal Definition of Myocardial Infarction". Time to cardiovascular death, myocardial infarction, or stroke was defined as the time from randomization to the first occurrence of any component of the composite endpoint and was analyzed using Kaplan-Meier (KM) survival analysis. KM estimates of the percentage of participants with an event are reported. Participants with no event were censored based on last non-fatal potential endpoint collection date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13447 | 13499
  KM estimate at 6 months | 1.86 [1.63 to 2.08] | 1.65 [1.44 to 1.86]
  KM estimate at 12 months: number analyzed (Participants) | 13140 | 13240
  KM estimate at 12 months | 3.68 [3.36 to 3.99] | 3.10 [2.81 to 3.38]
  KM estimate at 18 months: number analyzed (Participants) | 12257 | 12422
  KM estimate at 18 months | 5.18 [4.81 to 5.55] | 4.29 [3.95 to 4.62]
  KM estimate at 24 months: number analyzed (Participants) | 7923 | 8066
  KM estimate at 24 months | 6.83 [6.39 to 7.26] | 5.47 [5.08 to 5.86]
  KM estimate at 30 months: number analyzed (Participants) | 3785 | 3837
  KM estimate at 30 months | 8.31 [7.78 to 8.84] | 6.66 [6.19 to 7.14]
  KM estimate at 36 months: number analyzed (Participants) | 717 | 713
  KM estimate at 36 months | 9.93 [9.16 to 10.69] | 7.90 [7.17 to 8.63]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; If the primary endpoint reached statistical significance at the 0.05 level, the key secondary endpoint (composite of cardiovascular death, myocardial infarction, and stroke) was tested at a significance level of 0.05; Test type: Superiority; p < 0.0001, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.73 to 0.88] — Based on a Cox model stratified by the randomization stratification factors

3. Secondary Outcome: Time to Cardiovascular Death
Description: All deaths and potential endpoint events were adjudicated by an independent external CEC led by the TIMI Study Group, using standardized definitions based on the "Standardized Definitions for Cardiovascular and Stroke End Point Events in Clinical Trials and the Third Universal Definition of Myocardial Infarction".
  Cardiovascular death includes death resulting from an acute myocardial infarction (MI), sudden cardiac death, death due to heart failure (HF), death due to stroke, death due to cardiovascular (CV) procedures, death due to CV hemorrhage, and death due to other CV causes.
  Time to cardiovascular death was defined as the time from randomization to the date of cardiovascular death and was analyzed using Kaplan-Meier (KM) survival analysis. KM estimates of the percentage of participants with an event are reported. Participants with no event were censored based on the last confirmed survival status date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13688 | 13698
  KM estimate at 6 months | 0.40 [0.29 to 0.50] | 0.39 [0.29 to 0.50]
  KM estimate at 12 months: number analyzed (Participants) | 13590 | 13598
  KM estimate at 12 months | 0.82 [0.67 to 0.97] | 0.79 [0.64 to 0.94]
  KM estimate at 18 months: number analyzed (Participants) | 12844 | 12869
  KM estimate at 18 months | 1.19 [1.01 to 1.37] | 1.20 [1.01 to 1.38]
  KM estimate at 24 months: number analyzed (Participants) | 8427 | 8441
  KM estimate at 24 months | 1.57 [1.36 to 1.79] | 1.64 [1.42 to 1.85]
  KM estimate at 30 months: number analyzed (Participants) | 4081 | 4043
  KM estimate at 30 months | 1.99 [1.72 to 2.26] | 2.11 [1.83 to 2.39]
  KM estimate at 36 months: number analyzed (Participants) | 783 | 767
  KM estimate at 36 months | 2.39 [1.98 to 2.80] | 2.49 [2.09 to 2.88]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; If the primary and key secondary endpoints reached a statistical significance level of 0.05, then the endpoint of cardiovascular death was tested at a significance level of 0.05; Test type: Superiority; p = 0.6188, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.88 to 1.25] — Based on a Cox model stratified by the randomization stratification factors

4. Secondary Outcome: Time to All Cause Death
Description: Time to all-cause death was defined as the time from randomization to the date of death and was analyzed using Kaplan-Meier (KM) survival analysis. KM estimates of the percentage of participants with an event are reported. Participants with no event were censored based on the last confirmed survival status date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13688 | 13698
  KM estimate at 6 months | 0.62 [0.49 to 0.75] | 0.55 [0.43 to 0.68]
  KM estimate at 12 months: number analyzed (Participants) | 13590 | 13598
  KM estimate at 12 months | 1.29 [1.10 to 1.47] | 1.26 [1.07 to 1.44]
  KM estimate at 18 months: number analyzed (Participants) | 12844 | 12869
  KM estimate at 18 months | 1.96 [1.73 to 2.19] | 1.94 [1.71 to 2.17]
  KM estimate at 24 months: number analyzed (Participants) | 8427 | 8441
  KM estimate at 24 months | 2.78 [2.49 to 3.06] | 2.81 [2.52 to 3.10]
  KM estimate at 30 months: number analyzed (Participants) | 4081 | 4043
  KM estimate at 30 months | 3.48 [3.12 to 3.83] | 3.63 [3.27 to 3.98]
  KM estimate at 36 months: number analyzed (Participants) | 783 | 767
  KM estimate at 36 months | 4.28 [3.74 to 4.82] | 4.75 [4.16 to 5.34]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; If the primary, key secondary, and endpoint cardiovascular death reached a statistical significance level of 0.05, then the endpoint of all-cause death was tested at a significance level of 0.04 and remaining secondary endpoints at an overall significant level of 0.01 by applying the Hochberg method; Test type: Superiority; p = 0.5368, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.91 to 1.19] — Based on a Cox model stratified by the randomization stratification factors

5. Secondary Outcome: Time to First Myocardial Infarction
Description: All deaths and potential endpoint events were adjudicated by an independent external CEC led by the TIMI Study Group, using standardized definitions based on the "Standardized Definitions for Cardiovascular and Stroke End Point Events in Clinical Trials and the Third Universal Definition of Myocardial Infarction".
  The diagnosis of myocardial infarction required the combination of:
  * Evidence of myocardial necrosis (either changes in cardiac biomarkers or post-mortem pathological findings); and
  * Supporting information derived from the clinical presentation, electrocardiographic changes, or the results of myocardial or coronary artery Imaging.
  Time to first myocardial infarction was defined as the time from randomization to the date of the first MI and was analyzed using Kaplan-Meier survival analysis. KM estimates of the percentage of participants with an event are reported. Participants with no event were censored based on last non-fatal potential endpoint collection date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13497 | 13536
  KM estimate at 6 months | 1.14 [0.97 to 1.32] | 1.06 [0.88 to 1.23]
  KM estimate at 12 months: number analyzed (Participants) | 13226 | 13312
  KM estimate at 12 months | 2.39 [2.13 to 2.64] | 1.90 [1.67 to 2.13]
  KM estimate at 18 months: number analyzed (Participants) | 12374 | 12522
  KM estimate at 18 months | 3.33 [3.03 to 3.63] | 2.55 [2.28 to 2.81]
  KM estimate at 24 months: number analyzed (Participants) | 8031 | 8137
  KM estimate at 24 months | 4.30 [3.95 to 4.65] | 3.21 [2.90 to 3.51]
  KM estimate at 30 months: number analyzed (Participants) | 3839 | 3883
  KM estimate at 30 months | 5.25 [4.82 to 5.67] | 3.83 [3.47 to 4.19]
  KM estimate at 36 months: number analyzed (Participants) | 733 | 726
  KM estimate at 36 months | 6.28 [5.67 to 6.89] | 4.41 [3.85 to 4.96]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; If the primary, key secondary, and endpoint of cardiovascular death reached a statistical significance level of 0.05, then the endpoint of all-cause death was tested at a significance level of 0.04 and remaining secondary endpoints were tested at an overall significance level of 0.01 by applying the Hochberg method; Test type: Superiority; p < 0.0001, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.65 to 0.82] — Based on a Cox model stratified by the randomization stratification factors

6. Secondary Outcome: Time to First Stroke
Description: All deaths and potential endpoint events were adjudicated by an independent external CEC led by the TIMI Study Group, using standardized definitions based on the "Standardized Definitions for Cardiovascular and Stroke End Point Events in Clinical Trials and the Third Universal Definition of Myocardial Infarction".
  Stroke was defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction.
  Time to first stroke was defined as the time from randomization to the date of the stroke and was analyzed using Kaplan-Meier (KM) survival analysis. KM estimates of the percentage of participants with an event are reported. Participants with no event were censored based on last non-fatal potential endpoint collection date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13587 | 13631
  KM estimate at 6 months | 0.50 [0.38 to 0.61] | 0.31 [0.22 to 0.41]
  KM estimate at 12 months: number analyzed (Participants) | 13428 | 13470
  KM estimate at 12 months | 0.85 [0.69 to 1.00] | 0.70 [0.56 to 0.84]
  KM estimate at 18 months: number analyzed (Participants) | 12626 | 12703
  KM estimate at 18 months | 1.30 [1.11 to 1.50] | 1.05 [0.88 to 1.22]
  KM estimate at 24 months: number analyzed (Participants) | 8240 | 8304
  KM estimate at 24 months | 1.80 [1.57 to 2.04] | 1.36 [1.16 to 1.56]
  KM estimate at 30 months: number analyzed (Participants) | 3977 | 3967
  KM estimate at 30 months | 2.15 [1.88 to 2.43] | 1.71 [1.46 to 1.96]
  KM estimate at 36 months: number analyzed (Participants) | 757 | 741
  KM estimate at 36 months | 2.60 [2.20 to 3.00] | 2.18 [1.76 to 2.59]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0101, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.66 to 0.95] — Based on a Cox model stratified by the randomization stratification factors

7. Secondary Outcome: Time to First Coronary Revascularization
Description: All deaths and potential endpoint events were adjudicated by an independent external CEC led by the TIMI Study Group, using standardized definitions based on the "Standardized Definitions for Cardiovascular and Stroke End Point Events in Clinical Trials and the Third Universal Definition of Myocardial Infarction".
  Time to first coronary revascularization was defined as the time from randomization to the date of the coronary revascularization and was analyzed using Kaplan-Meier (KM) survival analysis. KM estimates of the percentage of participants with an event are reported. Participants with no event were censored based on last non-fatal potential endpoint collection date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13390 | 13454
  KM estimate at 6 months | 1.87 [1.65 to 2.10] | 1.60 [1.39 to 1.81]
  KM estimate at 12 months: number analyzed (Participants) | 13029 | 13130
  KM estimate at 12 months | 3.71 [3.39 to 4.02] | 3.13 [2.84 to 3.42]
  KM estimate at 18 months: number analyzed (Participants) | 12097 | 12283
  KM estimate at 18 months | 5.20 [4.82 to 5.57] | 4.16 [3.83 to 4.50]
  KM estimate at 24 months: number analyzed (Participants) | 7812 | 7952
  KM estimate at 24 months | 6.57 [6.14 to 7.00] | 5.22 [4.84 to 5.61]
  KM estimate at 30 months: number analyzed (Participants) | 3718 | 3768
  KM estimate at 30 months | 7.91 [7.39 to 8.42] | 6.13 [5.68 to 6.58]
  KM estimate at 36 months: number analyzed (Participants) | 704 | 710
  KM estimate at 36 months | 9.17 [8.46 to 9.87] | 7.01 [6.36 to 7.65]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.71 to 0.86] — Based on a Cox model stratified by the randomization stratification factors

8. Secondary Outcome: Time to Cardiovascular Death or First Hospitalization for Worsening Heart Failure
Description: All events were adjudicated by an independent external CEC led by the TIMI Study Group, using standardized definitions.
  HF hospitalization was defined as an event that met all of the following criteria:
  1. Admitted to hospital with a primary diagnosis of HF
  2. In hospital for at least 24 hours
  3. Documented new or worsening symptoms due to HF, including at least 1 of the following:
     * Dyspnea
     * Decreased exercise tolerance
     * Fatigue
     * Other symptoms of worsened end-organ perfusion or volume overload
  4. Evidence of new or worsening HF consisting of at least 2 physical exam findings or 1 physical exam finding and at least 1 laboratory criterion
  5. Received new or increased treatment for HF. Time to CV death or first hospitalization for worsening HF was defined as the time from randomization to the first occurrence of any component of the endpoint analyzed using KM survival analysis. Participants with no event were censored based on last non-fatal potential endpoint collection date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13592 | 13635
  KM estimate at 6 months | 0.79 [0.64 to 0.93] | 0.64 [0.51 to 0.77]
  KM estimate at 12 months: number analyzed (Participants) | 13455 | 13481
  KM estimate at 12 months | 1.35 [1.16 to 1.54] | 1.29 [1.10 to 1.48]
  KM estimate at 18 months: number analyzed (Participants) | 12664 | 12710
  KM estimate at 18 months | 1.99 [1.75 to 2.22] | 1.99 [1.76 to 2.22]
  KM estimate at 24 months: number analyzed (Participants) | 8265 | 8304
  KM estimate at 24 months | 2.70 [2.41 to 2.98] | 2.64 [2.36 to 2.92]
  KM estimate at 30 months: number analyzed (Participants) | 3983 | 3967
  KM estimate at 30 months | 3.45 [3.09 to 3.81] | 3.31 [2.97 to 3.65]
  KM estimate at 36 months: number analyzed (Participants) | 761 | 737
  KM estimate at 36 months | 4.03 [3.50 to 4.55] | 4.13 [3.57 to 4.68]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.8179, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.86 to 1.13] — Based on a Cox model stratified by the randomization stratification factors

9. Secondary Outcome: Time to First Ischemic Fatal or Non-Fatal Stroke or Transient Ischemic Attack
Description: All deaths and potential endpoint events were adjudicated by an independent external CEC led by the TIMI Study Group, using standardized definitions.
  Ischemic stroke was defined as an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of central nervous system tissue. Transient ischemic attack (TIA) was defined as a transient episode of focal neurological dysfunction caused by brain, spinal cord, or retinal ischemia, without acute infarction.
  Time to first ischemic fatal or non-fatal stroke or TIA was defined as the time from randomization to the first occurrence of any component of the composite endpoint and was analyzed using KM analysis. KM estimates of the percentage of participants with an event are reported. Participants with no event were censored based on last non-fatal potential endpoint collection date.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 13780 | 13784
percentage of participants
  KM estimate at 6 months: number analyzed (Participants) | 13569 | 13614
  KM estimate at 6 months | 0.61 [0.48 to 0.73] | 0.42 [0.31 to 0.53]
  KM estimate at 12 months: number analyzed (Participants) | 13394 | 13445
  KM estimate at 12 months | 1.05 [0.88 to 1.22] | 0.83 [0.67 to 0.98]
  KM estimate at 18 months: number analyzed (Participants) | 12588 | 12671
  KM estimate at 18 months | 1.52 [1.32 to 1.73] | 1.18 [1.00 to 1.37]
  KM estimate at 24 months: number analyzed (Participants) | 8209 | 8279
  KM estimate at 24 months | 2.05 [1.81 to 2.30] | 1.46 [1.25 to 1.66]
  KM estimate at 30 months: number analyzed (Participants) | 3958 | 3954
  KM estimate at 30 months | 2.40 [2.11 to 2.68] | 1.92 [1.65 to 2.19]
  KM estimate at 36 months: number analyzed (Participants) | 756 | 738
  KM estimate at 36 months | 2.81 [2.41 to 3.21] | 2.48 [2.01 to 2.95]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0035, Log Rank; Two-sided log-rank test stratified by randomization stratification factors (final screening LDL-C level and region); Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.65 to 0.92] — Based on a Cox model stratified by the randomization stratification factors

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to the end of study. The median duration of follow-up was 26 months.
Description: Deaths by any cause were adjudicated efficacy endpoints in this study and were summarized as a secondary endpoint. Events that were negatively adjudicated (did not meet the definitions of an endpoint), were reclassified as an adverse event or serious adverse event Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Evolocumab
Serious Adverse Events (participants affected / at risk) | 3404/13756 | 3410/13769
Other Adverse Events (participants affected / at risk) | 3438/13756 | 3500/13769
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13756) | Evolocumab (N=13769)
Anaemia (Blood and lymphatic system disorders) | 27 | 27
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 5 | 2
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 2
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 | 9
Leukocytosis (Blood and lymphatic system disorders) | 4 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 2
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 2 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 4
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 2
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 11 | 6
Acute left ventricular failure (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 23 | 11
Angina pectoris (Cardiac disorders) | 221 | 208
Angina unstable (Cardiac disorders) | 278 | 233
Aortic valve disease (Cardiac disorders) | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 2 | 2
Aortic valve stenosis (Cardiac disorders) | 8 | 10
Arrhythmia (Cardiac disorders) | 4 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 3
Arteritis coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 132 | 119
Atrial flutter (Cardiac disorders) | 17 | 25
Atrial tachycardia (Cardiac disorders) | 2 | 2
Atrial thrombosis (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 5 | 4
Atrioventricular block complete (Cardiac disorders) | 13 | 16
Atrioventricular block first degree (Cardiac disorders) | 3 | 1
Atrioventricular block second degree (Cardiac disorders) | 7 | 7
Bifascicular block (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 13 | 10
Bundle branch block bilateral (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 3
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac aneurysm (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 5 | 3
Cardiac asthma (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 66 | 66
Cardiac failure acute (Cardiac disorders) | 10 | 13
Cardiac failure chronic (Cardiac disorders) | 47 | 50
Cardiac failure congestive (Cardiac disorders) | 37 | 46
Cardiac flutter (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 3 | 2
Cardiomyopathy (Cardiac disorders) | 4 | 2
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 1 | 0
Cardiotoxicity (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 46 | 32
Coronary artery occlusion (Cardiac disorders) | 4 | 1
Coronary artery stenosis (Cardiac disorders) | 4 | 5
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Dressler's syndrome (Cardiac disorders) | 1 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Heart alternation (Cardiac disorders) | 1 | 0
Heart valve incompetence (Cardiac disorders) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 6 | 7
Left ventricular dysfunction (Cardiac disorders) | 7 | 1
Left ventricular failure (Cardiac disorders) | 2 | 1
Microvascular coronary artery disease (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 3 | 11
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 31 | 31
Myocardial ischaemia (Cardiac disorders) | 21 | 26
Myocardial necrosis (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 2 | 1
Palpitations (Cardiac disorders) | 8 | 7
Pericardial effusion (Cardiac disorders) | 2 | 3
Pericarditis (Cardiac disorders) | 2 | 4
Prinzmetal angina (Cardiac disorders) | 3 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Rhythm idioventricular (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 2 | 1
Sinus arrest (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 4 | 4
Sinus node dysfunction (Cardiac disorders) | 18 | 17
Sinus tachycardia (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 9 | 9
Tachycardia (Cardiac disorders) | 4 | 3
Torsade de pointes (Cardiac disorders) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 6 | 4
Ventricular extrasystoles (Cardiac disorders) | 5 | 7
Ventricular fibrillation (Cardiac disorders) | 8 | 12
Ventricular hypertrophy (Cardiac disorders) | 0 | 1
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 27 | 23
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 2
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 2 | 0
Carbohydrate metabolism disorder (Congenital, familial and genetic disorders) | 2 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 1
Exomphalos (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Hereditary motor and sensory neuropathy (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 2
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Intracranial lipoma (Congenital, familial and genetic disorders) | 1 | 0
Subependymal nodular heterotopia (Congenital, familial and genetic disorders) | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 2
Deafness (Ear and labyrinth disorders) | 1 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Inner ear inflammation (Ear and labyrinth disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 2
Otorrhoea (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 13 | 9
Vertigo positional (Ear and labyrinth disorders) | 1 | 7
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Vestibular ischaemia (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 1
Adrenal mass (Endocrine disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 3 | 3
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 3 | 4
Hypoaldosteronism (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 4 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1
Blepharochalasis (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 22 | 15
Cataract nuclear (Eye disorders) | 1 | 0
Dacryoadenitis acquired (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 2
Ectropion (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 2 | 1
Glaucoma (Eye disorders) | 1 | 1
Iridocyclitis (Eye disorders) | 1 | 1
Macular degeneration (Eye disorders) | 1 | 1
Macular fibrosis (Eye disorders) | 1 | 3
Ocular myasthenia (Eye disorders) | 0 | 1
Ophthalmoplegia (Eye disorders) | 0 | 1
Pterygium (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal artery thrombosis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 5 | 3
Retinal tear (Eye disorders) | 0 | 1
Retinal vascular disorder (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 1
Uveitis (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 2
Abdominal adhesions (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal hernia (Gastrointestinal disorders) | 8 | 11
Abdominal pain (Gastrointestinal disorders) | 19 | 12
Abdominal pain lower (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 13 | 12
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 2
Alcoholic pancreatitis (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 2
Anal fistula (Gastrointestinal disorders) | 4 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1
Anastomotic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 3 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 2 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 3
Coeliac artery stenosis (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 8 | 6
Colitis ischaemic (Gastrointestinal disorders) | 2 | 10
Colitis ulcerative (Gastrointestinal disorders) | 5 | 2
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 9
Crohn's disease (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 9
Diverticulum (Gastrointestinal disorders) | 4 | 4
Diverticulum intestinal (Gastrointestinal disorders) | 3 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 4 | 1
Duodenal ulcer (Gastrointestinal disorders) | 5 | 5
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 5 | 5
Duodenitis (Gastrointestinal disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 7
Dysphagia (Gastrointestinal disorders) | 4 | 1
Enteritis (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 2
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 4
Food poisoning (Gastrointestinal disorders) | 1 | 4
Gastric cyst (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 8 | 9
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 6 | 7
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 17 | 19
Gastritis alcoholic (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 3 | 3
Gastritis haemorrhagic (Gastrointestinal disorders) | 3 | 0
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 2
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 16 | 27
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 | 14
Haematemesis (Gastrointestinal disorders) | 2 | 4
Haematochezia (Gastrointestinal disorders) | 1 | 4
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 5 | 3
Haemorrhoids (Gastrointestinal disorders) | 10 | 6
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 3 | 9
Ileus (Gastrointestinal disorders) | 7 | 6
Ileus paralytic (Gastrointestinal disorders) | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 3
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 22 | 32
Intestinal dilatation (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 3
Intestinal polyp (Gastrointestinal disorders) | 2 | 1
Intestinal prolapse (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 16 | 10
Leukoplakia oral (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 2 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 1
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 5
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 1
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 3 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 2 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 4 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Palatal swelling (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 2 | 0
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatic phlegmon (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 16 | 10
Pancreatitis acute (Gastrointestinal disorders) | 22 | 14
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 3
Pancreatolithiasis (Gastrointestinal disorders) | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Peritoneal haematoma (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 9 | 6
Rectal polyp (Gastrointestinal disorders) | 2 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 6 | 4
Small intestine ulcer (Gastrointestinal disorders) | 1 | 0
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 | 1
Stress ulcer (Gastrointestinal disorders) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1
Tongue cyst (Gastrointestinal disorders) | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 14 | 10
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 13
Varices oesophageal (Gastrointestinal disorders) | 1 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 4
Asthenia (General disorders) | 6 | 8
Breakthrough pain (General disorders) | 1 | 0
Catheter site extravasation (General disorders) | 1 | 0
Chest discomfort (General disorders) | 5 | 4
Chest pain (General disorders) | 49 | 42
Complication associated with device (General disorders) | 0 | 2
Cyst rupture (General disorders) | 0 | 1
Drug intolerance (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 2
Fat necrosis (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 2
Gait disturbance (General disorders) | 0 | 5
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 2
Impaired healing (General disorders) | 5 | 4
Implant site inflammation (General disorders) | 0 | 1
Incarcerated hernia (General disorders) | 0 | 2
Inflammation (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 3
Mass (General disorders) | 0 | 1
Medical device discomfort (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 133 | 109
Oedema peripheral (General disorders) | 1 | 4
Pacemaker generated arrhythmia (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 9 | 5
Sensation of foreign body (General disorders) | 1 | 0
Soft tissue inflammation (General disorders) | 0 | 1
Strangulated hernia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Surgical failure (General disorders) | 2 | 0
Systemic inflammatory response syndrome (General disorders) | 3 | 1
Vascular stent occlusion (General disorders) | 1 | 1
Vascular stent restenosis (General disorders) | 1 | 2
Vascular stent stenosis (General disorders) | 3 | 2
Vascular stent thrombosis (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 1
Ampulla of Vater stenosis (Hepatobiliary disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 5 | 6
Biliary colic (Hepatobiliary disorders) | 5 | 4
Biliary cyst (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 5
Cholangitis acute (Hepatobiliary disorders) | 6 | 0
Cholecystitis (Hepatobiliary disorders) | 7 | 14
Cholecystitis acute (Hepatobiliary disorders) | 31 | 40
Cholecystitis chronic (Hepatobiliary disorders) | 5 | 5
Cholecystocholangitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 23 | 27
Cholelithiasis migration (Hepatobiliary disorders) | 1 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 3
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Porcelain gallbladder (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 1
Subacute hepatic failure (Hepatobiliary disorders) | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 3 | 2
Anaphylactic shock (Immune system disorders) | 0 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 1
Mite allergy (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess bacterial (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 4 | 10
Abscess of eyelid (Infections and infestations) | 0 | 1
Abscess of salivary gland (Infections and infestations) | 0 | 1
Abscess soft tissue (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 5 | 2
Anal fistula infection (Infections and infestations) | 1 | 0
Appendiceal abscess (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 14 | 20
Appendicitis perforated (Infections and infestations) | 5 | 2
Arteritis infective (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 2 | 0
Atypical pneumonia (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial pericarditis (Infections and infestations) | 0 | 1
Bacterial prostatitis (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bacteroides bacteraemia (Infections and infestations) | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Bone abscess (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 30 | 17
Bronchitis bacterial (Infections and infestations) | 2 | 2
Burkholderia cepacia complex infection (Infections and infestations) | 1 | 0
Burkholderia pseudomallei infection (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 2
Campylobacter gastroenteritis (Infections and infestations) | 1 | 2
Carbuncle (Infections and infestations) | 2 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 28 | 39
Cellulitis gangrenous (Infections and infestations) | 1 | 0
Cervicitis (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 2 | 2
Chronic hepatitis B (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 6
Clostridium difficile infection (Infections and infestations) | 2 | 3
Colonic abscess (Infections and infestations) | 0 | 1
Creutzfeldt-Jakob disease (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 5 | 3
Cystitis escherichia (Infections and infestations) | 1 | 1
Dengue fever (Infections and infestations) | 4 | 1
Device related infection (Infections and infestations) | 3 | 1
Device related sepsis (Infections and infestations) | 1 | 2
Diabetic foot infection (Infections and infestations) | 6 | 2
Diabetic gangrene (Infections and infestations) | 1 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 26 | 16
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 1
Eczema infected (Infections and infestations) | 1 | 0
Embolic pneumonia (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 3 | 0
Encephalitis viral (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Endocarditis haemophilus (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 2 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 3 | 1
Epiglottitis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 19 | 16
Erysipeloid (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 3 | 4
Escherichia urinary tract infection (Infections and infestations) | 0 | 2
Febrile infection (Infections and infestations) | 0 | 1
Fungal peritonitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 12 | 6
Gastritis viral (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 14 | 19
Gastroenteritis adenovirus (Infections and infestations) | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 2
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 1 | 1
Gastroenteritis salmonella (Infections and infestations) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 3 | 3
Gastrointestinal infection (Infections and infestations) | 2 | 1
Gingival abscess (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 2 | 1
Groin abscess (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 2 | 1
Hepatitis C (Infections and infestations) | 0 | 3
Hepatitis E (Infections and infestations) | 1 | 3
Herpes zoster (Infections and infestations) | 3 | 5
Implant site infection (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Infected bite (Infections and infestations) | 1 | 1
Infected cyst (Infections and infestations) | 3 | 0
Infected skin ulcer (Infections and infestations) | 2 | 2
Infection (Infections and infestations) | 0 | 1
Infection in an immunocompromised host (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 2 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 5 | 3
Infective tenosynovitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 6 | 9
Intervertebral discitis (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 1
Laryngitis (Infections and infestations) | 2 | 1
Liver abscess (Infections and infestations) | 0 | 2
Localised infection (Infections and infestations) | 6 | 6
Lower respiratory tract infection (Infections and infestations) | 15 | 14
Lower respiratory tract infection viral (Infections and infestations) | 0 | 2
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 5
Mastoiditis (Infections and infestations) | 1 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Medical device site infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Meningitis pneumococcal (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 2
Neurosyphilis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 1
Oral fungal infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 2 | 2
Osteomyelitis (Infections and infestations) | 7 | 16
Osteomyelitis acute (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 2 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis externa bacterial (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 2
Pancreas infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 2 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 2 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 2 | 4
Peritonitis bacterial (Infections and infestations) | 2 | 1
Pharyngeal abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 152 | 147
Pneumonia adenoviral (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 11 | 18
Pneumonia influenzal (Infections and infestations) | 1 | 1
Pneumonia legionella (Infections and infestations) | 1 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 3 | 4
Post procedural pneumonia (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 1 | 1
Postoperative abscess (Infections and infestations) | 4 | 0
Postoperative wound infection (Infections and infestations) | 8 | 3
Prostate infection (Infections and infestations) | 0 | 1
Prostatic abscess (Infections and infestations) | 1 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 1
Psoas abscess (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 3 | 0
Pyelonephritis (Infections and infestations) | 4 | 10
Pyelonephritis acute (Infections and infestations) | 6 | 6
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Pyonephrosis (Infections and infestations) | 1 | 1
Rectal abscess (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 8 | 8
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Salpingitis (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 1
Scrotal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 31 | 21
Septic shock (Infections and infestations) | 9 | 6
Sinusitis (Infections and infestations) | 1 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 2 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Spermatic cord funiculitis (Infections and infestations) | 0 | 1
Splenic abscess (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 3 | 1
Staphylococcal infection (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 2 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 2
Testicular abscess (Infections and infestations) | 0 | 1
Tick-borne viral encephalitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 3
Tracheitis (Infections and infestations) | 0 | 2
Tracheobronchitis (Infections and infestations) | 3 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 6
Upper respiratory tract infection bacterial (Infections and infestations) | 3 | 0
Ureteritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 37 | 41
Urinary tract infection bacterial (Infections and infestations) | 7 | 7
Urosepsis (Infections and infestations) | 15 | 12
Vestibular neuronitis (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 3 | 4
Viral myocarditis (Infections and infestations) | 1 | 0
Viral pericarditis (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 2
Wound abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 11 | 6
Wound infection bacterial (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 2 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 3
Acetabulum fracture (Injury, poisoning and procedural complications) | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 | 3
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic fistula (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 2
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 12 | 8
Aortic injury (Injury, poisoning and procedural complications) | 0 | 1
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 | 1
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Arterial restenosis (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 2
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 4
Chemical burn of gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 3
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 3 | 5
Contusion (Injury, poisoning and procedural complications) | 3 | 6
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 2
Cranial nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 | 6
Diffuse axonal injury (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of sternum (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 2 | 1
Eye operation complication (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 4 | 3
Fall (Injury, poisoning and procedural complications) | 13 | 17
Femoral neck fracture (Injury, poisoning and procedural complications) | 7 | 4
Femur fracture (Injury, poisoning and procedural complications) | 9 | 20
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 4 | 5
Forearm fracture (Injury, poisoning and procedural complications) | 3 | 4
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Graft complication (Injury, poisoning and procedural complications) | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 3 | 0
Head injury (Injury, poisoning and procedural complications) | 8 | 6
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 11 | 11
Humerus fracture (Injury, poisoning and procedural complications) | 8 | 6
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 4 | 5
Incomplete spinal fusion (Injury, poisoning and procedural complications) | 0 | 1
Inflammation of wound (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 5
Intentional overdose (Injury, poisoning and procedural complications) | 5 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 5 | 4
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 2
Kidney contusion (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 4 | 4
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 3
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 1
Limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 3 | 2
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 4
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 | 7
Medication error (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 4 | 8
Metal poisoning (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Open globe injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 2
Patella fracture (Injury, poisoning and procedural complications) | 3 | 4
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 1
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 0 | 2
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 2 | 2
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Peroneal nerve palsy postoperative (Injury, poisoning and procedural complications) | 0 | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 | 1
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 1
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 1
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 2
Post procedural constipation (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 | 3
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 7 | 6
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 2 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 2 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2
Procedural pneumothorax (Injury, poisoning and procedural complications) | 3 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 2 | 2
Radial head dislocation (Injury, poisoning and procedural complications) | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 4 | 1
Rib fracture (Injury, poisoning and procedural complications) | 11 | 7
Road traffic accident (Injury, poisoning and procedural complications) | 6 | 4
Sacroiliac fracture (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 3 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 3
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 2
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 5
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury lumbar (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 3 | 2
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 2 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 3 | 3
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 11 | 6
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 3
Tendon injury (Injury, poisoning and procedural complications) | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 8 | 6
Thermal burn (Injury, poisoning and procedural complications) | 2 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 7
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 2
Traumatic haemothorax (Injury, poisoning and procedural complications) | 3 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Traumatic shock (Injury, poisoning and procedural complications) | 0 | 1
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 5
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 0 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 2 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 5 | 2
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 3
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 | 2
Wound (Injury, poisoning and procedural complications) | 3 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 4
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 3
Alanine aminotransferase increased (Investigations) | 15 | 11
Arteriogram coronary (Investigations) | 3 | 5
Arteriogram coronary abnormal (Investigations) | 2 | 1
Arteriogram coronary normal (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 11 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 6 | 7
Blood creatinine increased (Investigations) | 1 | 2
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose fluctuation (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 2
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Cardiac stress test abnormal (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 2 | 4
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 2
Electrocardiogram abnormal (Investigations) | 1 | 1
Exercise electrocardiogram abnormal (Investigations) | 0 | 1
False positive investigation result (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 8 | 24
Hepatitis A antibody positive (Investigations) | 0 | 1
Hepatitis A virus test positive (Investigations) | 0 | 1
Hepatitis B antibody positive (Investigations) | 1 | 0
Hepatitis C virus test positive (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 1
Influenza B virus test positive (Investigations) | 0 | 1
International normalised ratio abnormal (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 4 | 1
Investigation (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 4 | 7
Liver function test increased (Investigations) | 7 | 0
Medical observation (Investigations) | 0 | 1
Myocardial necrosis marker increased (Investigations) | 1 | 2
Oxygen saturation decreased (Investigations) | 1 | 0
Precancerous cells present (Investigations) | 1 | 0
Stress echocardiogram (Investigations) | 0 | 1
Thyroid function test abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 5 | 6
Troponin I increased (Investigations) | 2 | 1
Troponin T increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 2 | 3
Weight decreased (Investigations) | 2 | 0
Weight increased (Investigations) | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 18 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 56 | 61
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 11 | 6
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 8 | 10
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 3 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 3
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 5 | 6
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 8
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 10
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 17
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 5
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 2
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 2
Obesity (Metabolism and nutrition disorders) | 6 | 3
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 12
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 13 | 11
Arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 30
Bone deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 3
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 5 | 7
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 | 8
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 4
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 24 | 22
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint adhesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 17 | 21
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 37 | 49
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 | 2
Myofascitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 100 | 91
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 2
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 7 | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 9 | 8
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 5 | 6
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 9
Spinal pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 3
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 5 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 17
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 4
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Biliary adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 12
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder cancer stage I, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 9
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 11
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Endometrial adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Gastric cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Large cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lip and/or oral cavity cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 13
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung carcinoma cell type unspecified stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 19
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung squamous cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma of sites other than skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Oral cavity cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pharyngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 40 | 41
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Rectal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 9
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Small cell lung cancer limited stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Undifferentiated sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vulval cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 4 | 2
Amnesia (Nervous system disorders) | 0 | 2
Amputation stump pain (Nervous system disorders) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 2 | 0
Apraxia (Nervous system disorders) | 1 | 0
Arachnoid cyst (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 1
Basal ganglia infarction (Nervous system disorders) | 0 | 1
Basilar artery aneurysm (Nervous system disorders) | 0 | 1
Basilar artery stenosis (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 6 | 5
Carotid artery disease (Nervous system disorders) | 2 | 3
Carotid artery occlusion (Nervous system disorders) | 7 | 3
Carotid artery stenosis (Nervous system disorders) | 39 | 37
Carpal tunnel syndrome (Nervous system disorders) | 3 | 6
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cerebellar ataxia (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebral artery occlusion (Nervous system disorders) | 1 | 1
Cerebral artery stenosis (Nervous system disorders) | 0 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 3 | 5
Cerebral ischaemia (Nervous system disorders) | 6 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 1
Cerebral vasoconstriction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 21 | 25
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 2
Cervical cord compression (Nervous system disorders) | 0 | 1
Cervical myelopathy (Nervous system disorders) | 1 | 2
Cervical radiculopathy (Nervous system disorders) | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 3
Cervicogenic headache (Nervous system disorders) | 0 | 1
Complex partial seizures (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 6 | 4
Dizziness (Nervous system disorders) | 19 | 15
Dizziness postural (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 2
Dystonia (Nervous system disorders) | 1 | 0
Encephalitis autoimmune (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 2
Epilepsy (Nervous system disorders) | 7 | 5
Facial paralysis (Nervous system disorders) | 4 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 2 | 2
Guillain-Barre syndrome (Nervous system disorders) | 3 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 17 | 9
Hemiparesis (Nervous system disorders) | 1 | 4
Hemiplegic migraine (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 2 | 0
Hypertonia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 3
Hypoglycaemic coma (Nervous system disorders) | 3 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 | 0
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 6 | 3
Intracranial mass (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 2
Ischaemic stroke (Nervous system disorders) | 5 | 6
Lacunar infarction (Nervous system disorders) | 2 | 2
Lacunar stroke (Nervous system disorders) | 3 | 0
Lethargy (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 7 | 2
Lumbar radiculopathy (Nervous system disorders) | 1 | 3
Lumbosacral radiculopathy (Nervous system disorders) | 2 | 0
Meralgia paraesthetica (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 3 | 3
Migraine with aura (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 1 | 0
Motor neurone disease (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 2 | 1
Nerve compression (Nervous system disorders) | 1 | 1
Nervous system disorder (Nervous system disorders) | 1 | 1
Neuralgia (Nervous system disorders) | 3 | 2
Neuritis (Nervous system disorders) | 1 | 0
Neuroglycopenia (Nervous system disorders) | 0 | 1
Neuromuscular pain (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 5
Paraesthesia (Nervous system disorders) | 4 | 3
Paraparesis (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 2 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 1
Petit mal epilepsy (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 2 | 0
Polyneuropathy idiopathic progressive (Nervous system disorders) | 1 | 0
Postictal state (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 4 | 9
Pseudoradicular syndrome (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Quadriplegia (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 2 | 6
Retrograde amnesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 10 | 14
Sedation (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 13 | 8
Speech disorder (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 2 | 0
Stroke in evolution (Nervous system disorders) | 2 | 1
Subdural effusion (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 56 | 63
Tarsal tunnel syndrome (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 0 | 3
Thoracic outlet syndrome (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 36 | 42
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 2 | 3
Vertebral artery occlusion (Nervous system disorders) | 0 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 5 | 4
Vertigo CNS origin (Nervous system disorders) | 0 | 2
Visual field defect (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Device battery issue (Product Issues) | 1 | 0
Device breakage (Product Issues) | 1 | 1
Device dislocation (Product Issues) | 2 | 1
Device failure (Product Issues) | 3 | 0
Device ineffective (Product Issues) | 0 | 1
Device leakage (Product Issues) | 0 | 1
Device loosening (Product Issues) | 1 | 1
Device malfunction (Product Issues) | 5 | 5
Device occlusion (Product Issues) | 3 | 1
Lead dislodgement (Product Issues) | 1 | 0
Thrombosis in device (Product Issues) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 4 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 3
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 7 | 4
Anxiety disorder (Psychiatric disorders) | 4 | 0
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Burnout syndrome (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 4
Conversion disorder (Psychiatric disorders) | 1 | 3
Delirium (Psychiatric disorders) | 3 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 20 | 15
Depression suicidal (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 2 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 4 | 1
Mania (Psychiatric disorders) | 1 | 2
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 4 | 6
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 | 1
Neurosis (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 3
Personality disorder (Psychiatric disorders) | 0 | 1
Psychiatric decompensation (Psychiatric disorders) | 0 | 1
Psychogenic seizure (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 3 | 1
Somatic symptom disorder (Psychiatric disorders) | 1 | 2
Suicidal ideation (Psychiatric disorders) | 3 | 3
Suicide attempt (Psychiatric disorders) | 6 | 6
Acute kidney injury (Renal and urinary disorders) | 64 | 64
Acute prerenal failure (Renal and urinary disorders) | 2 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Bladder dilatation (Renal and urinary disorders) | 1 | 0
Bladder diverticulum (Renal and urinary disorders) | 1 | 2
Bladder neck obstruction (Renal and urinary disorders) | 1 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 2 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 3
Calculus urinary (Renal and urinary disorders) | 6 | 3
Chronic kidney disease (Renal and urinary disorders) | 15 | 17
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 4 | 2
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 12 | 17
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 4 | 3
Nephrolithiasis (Renal and urinary disorders) | 29 | 16
Nephropathy toxic (Renal and urinary disorders) | 1 | 2
Nephrotic syndrome (Renal and urinary disorders) | 2 | 2
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 2
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 6 | 1
Renal colic (Renal and urinary disorders) | 4 | 3
Renal cyst (Renal and urinary disorders) | 0 | 2
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 5
Renal impairment (Renal and urinary disorders) | 4 | 4
Renal infarct (Renal and urinary disorders) | 0 | 2
Renal mass (Renal and urinary disorders) | 2 | 0
Renal pain (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 3
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 0
Ureteric rupture (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 5 | 9
Urethral stenosis (Renal and urinary disorders) | 4 | 5
Urinary incontinence (Renal and urinary disorders) | 6 | 1
Urinary retention (Renal and urinary disorders) | 4 | 14
Urinary tract obstruction (Renal and urinary disorders) | 3 | 3
Urinoma (Renal and urinary disorders) | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 26 | 30
Breast dysplasia (Reproductive system and breast disorders) | 0 | 1
Breast enlargement (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 1
Cervix disorder (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 2
Endometrial thickening (Reproductive system and breast disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 1
Male genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 3 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 5 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 1
Reproductive tract disorder (Reproductive system and breast disorders) | 0 | 1
Scrotal cyst (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Spermatic cord inflammation (Reproductive system and breast disorders) | 1 | 0
Uterine atony (Reproductive system and breast disorders) | 0 | 1
Uterine enlargement (Reproductive system and breast disorders) | 1 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 2 | 0
Uterine polyp (Reproductive system and breast disorders) | 2 | 2
Uterine prolapse (Reproductive system and breast disorders) | 0 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 3
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Vulval disorder (Reproductive system and breast disorders) | 1 | 0
Vulvar dysplasia (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 64 | 64
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 28
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural adhesion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 28 | 20
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 16
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 7 | 6
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0
Excessive skin (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen myxoedematosus (Skin and subcutaneous tissue disorders) | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Papulopustular rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 | 5
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3
Abstains from alcohol (Social circumstances) | 1 | 0
Disability (Social circumstances) | 1 | 0
Social stay hospitalisation (Social circumstances) | 0 | 1
Substance abuser (Social circumstances) | 1 | 0
Abscess drainage (Surgical and medical procedures) | 1 | 1
Aortic valve replacement (Surgical and medical procedures) | 1 | 0
Arrhythmia prophylaxis (Surgical and medical procedures) | 0 | 1
Arterial catheterisation (Surgical and medical procedures) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 1
Asthma prophylaxis (Surgical and medical procedures) | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 1
Cardiac rehabilitation therapy (Surgical and medical procedures) | 1 | 0
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 | 2
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Coronary revascularisation (Surgical and medical procedures) | 2 | 1
Elective procedure (Surgical and medical procedures) | 1 | 0
Enterostomy (Surgical and medical procedures) | 0 | 1
Finger amputation (Surgical and medical procedures) | 0 | 1
Fracture treatment (Surgical and medical procedures) | 1 | 0
Gastric banding reversal (Surgical and medical procedures) | 1 | 0
Haemostasis (Surgical and medical procedures) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 2 | 0
Incisional hernia repair (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 3
Knee arthroplasty (Surgical and medical procedures) | 0 | 3
Large intestinal polypectomy (Surgical and medical procedures) | 0 | 1
Large intestine anastomosis (Surgical and medical procedures) | 1 | 0
Leg amputation (Surgical and medical procedures) | 2 | 0
Open reduction of fracture (Surgical and medical procedures) | 0 | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 1 | 3
Peripheral artery bypass (Surgical and medical procedures) | 2 | 0
Plastic surgery to the face (Surgical and medical procedures) | 1 | 0
Preoperative care (Surgical and medical procedures) | 1 | 0
Proctectomy (Surgical and medical procedures) | 1 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 2
Spinal anaesthesia (Surgical and medical procedures) | 0 | 1
Stent placement (Surgical and medical procedures) | 0 | 1
Therapy cessation (Surgical and medical procedures) | 1 | 0
Toe amputation (Surgical and medical procedures) | 0 | 1
Transcatheter aortic valve implantation (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Umbilical hernia repair (Surgical and medical procedures) | 0 | 1
Urethral operation (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 2 | 3
Aneurysm (Vascular disorders) | 4 | 0
Angiopathy (Vascular disorders) | 1 | 0
Angiosclerosis (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 27 | 27
Aortic aneurysm rupture (Vascular disorders) | 1 | 1
Aortic occlusion (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 8 | 7
Aortic thrombosis (Vascular disorders) | 1 | 1
Arterial occlusive disease (Vascular disorders) | 5 | 1
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 4 | 2
Arteriovenous fistula (Vascular disorders) | 1 | 0
Blood pressure fluctuation (Vascular disorders) | 1 | 1
Circulatory collapse (Vascular disorders) | 6 | 5
Cryoglobulinaemia (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 14 | 7
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Dry gangrene (Vascular disorders) | 0 | 4
Embolism (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 2 | 0
Embolism venous (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 4 | 2
Granulomatosis with polyangiitis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 5 | 2
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 41 | 56
Hypertensive crisis (Vascular disorders) | 12 | 15
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 13 | 9
Hypovolaemic shock (Vascular disorders) | 2 | 1
Iliac artery occlusion (Vascular disorders) | 3 | 5
Intermittent claudication (Vascular disorders) | 22 | 31
Internal haemorrhage (Vascular disorders) | 1 | 0
Leriche syndrome (Vascular disorders) | 2 | 1
Lymphocele (Vascular disorders) | 1 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 2 | 1
Neurogenic shock (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 7 | 9
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 82 | 94
Peripheral artery aneurysm (Vascular disorders) | 7 | 5
Peripheral artery dissection (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 16 | 20
Peripheral artery stenosis (Vascular disorders) | 33 | 27
Peripheral artery thrombosis (Vascular disorders) | 5 | 5
Peripheral circulatory failure (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 3 | 1
Peripheral ischaemia (Vascular disorders) | 39 | 35
Peripheral vascular disorder (Vascular disorders) | 9 | 16
Peripheral venous disease (Vascular disorders) | 2 | 2
Poor peripheral circulation (Vascular disorders) | 1 | 0
Renovascular hypertension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 2 | 1
Subclavian artery embolism (Vascular disorders) | 1 | 0
Subclavian artery occlusion (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 5 | 4
Subclavian steal syndrome (Vascular disorders) | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Takayasu's arteritis (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 1 | 1
Thromboangiitis obliterans (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 2 | 2
Varicose ulceration (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 4 | 3
Vascular insufficiency (Vascular disorders) | 0 | 1
Vascular occlusion (Vascular disorders) | 0 | 1
Vascular stenosis (Vascular disorders) | 0 | 2
Vasodilatation (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13756) | Evolocumab (N=13769)
Nasopharyngitis (Infections and infestations) | 1021 | 1067
Upper respiratory tract infection (Infections and infestations) | 649 | 692
Diabetes mellitus (Metabolism and nutrition disorders) | 1096 | 1156
Hypertension (Vascular disorders) | 1157 | 1069

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.